CLINICAL TRIAL: NCT02978287
Title: The Effects of Cold Ischemia Time With a New Transporting Solution to Parathyroid Cell Viability and Calcium Sensing Receptor in Parathyroid Allotransplantation
Brief Title: New Transporting Solution in Parathyroid Allotransplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Principal Investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BAVU Solusyon
Record Dates: First submitted 2016-11-24; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Parathyroid Allotransplantation
Keywords: Calcium sensing receptor; Parathyroid cell viability; Parathyroid allotransplantation; Transporting solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- BAVU Solution 0. hour (control) (No Intervention): Viability, Calcium sensing receptor and parathormone levels of Parathyroid cells at 0. hour
- BAVU Solution 6. hour (Experimental): Viability, Calcium sensing receptor and parathormone levels of Parathyroid cells at 6. hour
  Interventions: Drug: BAVU Solution
- BAVU Solution 12. hour (Experimental): Viability, Calcium sensing receptor and parathormone levels of Parathyroid cells at 12. hour
  Interventions: Drug: BAVU Solution
- BAVU Solution 18. hour (Experimental): Viability, Calcium sensing receptor and parathormone levels of Parathyroid cells at 18. hour
  Interventions: Drug: BAVU Solution
- BAVU Solution 24. hour (Experimental): Viability, Calcium sensing receptor and parathormone levels of Parathyroid cells at 24. hour
  Interventions: Drug: BAVU Solution

INTERVENTIONS:
Drug: BAVU Solution — Tissue preservation solution for transplantation
  Arms: BAVU Solution 12. hour; BAVU Solution 18. hour; BAVU Solution 24. hour; BAVU Solution 6. hour

SUMMARY:
The aim of this study is to measure of the parathyroid cell viability and the the amount of calcium sensing receptor of the parathyroid cells which were placed into a new transportation solution (BAVU solution) for parathyroid allotransplantation.

DETAILED DESCRIPTION:
The cold ischemia of organs, has harmful effects on the tissues due to oxidative stress and inflammation. This is physiopathologically defined as ischaemia/re-perfusion injury (IRI) in organ transplantation. Parathyroid allotransplantation has an increased popularity at the last decade. But the cold ischemia due to transportation of the transplant tissue is a very important problem.

Calcium sensing receptor plays a crucial role in regulating Parathormone secretion which means controlling of the calcium-dependent systemic ion homeostasis.

The investigators developed a new tissue transporting solution for parathyroid allotransplantation and the investigators measured the parathyroid cell viability and the the amount of calcium sensing receptor of the parathyroid cells at the 0., 6., 12. and 24. hours of the parathyroid cells which were placed into our new solution.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have parathyroid hyperplasia due to chronic renal failure

Exclusion Criteria:

* Patients who refused to join to the study
* Patients younger than 18 years and older than 80 years.
* Patients who have hepatitis B,
* Patients who have hepatitis C,
* Patients who have human immunodeficiency virus (HIV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Cell viability of Parathyroid cells | 0 hour
  The investigators will measure the viability of Parathyroid cells at 0 hour at the BAVU solution
Cell viability of Parathyroid cells | 6 hours
  The investigators will measure the viability of Parathyroid cells at 6 hours at the BAVU solution
Cell viability of Parathyroid cells | 12 hours
  The investigators will measure the viability of Parathyroid cells at 12 hours at the BAVU solution
Cell viability of Parathyroid cells | 18 hours
  The investigators will measure the viability of Parathyroid cells at 18 hours at the BAVU solution
Cell viability of Parathyroid cells | 24 hours
  The investigators will measure the viability of Parathyroid cells at 24 hours at the BAVU solution

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guibert EE, Petrenko AY, Balaban CL, Somov AY, Rodriguez JV, Fuller BJ. Organ Preservation: Current Concepts and New Strategies for the Next Decade. Transfus Med Hemother. 2011;38(2):125-142. doi: 10.1159/000327033. Epub 2011 Mar 21. PMID 21566713
- [Result] Hendy GN, Guarnieri V, Canaff L. Calcium-sensing receptor and associated diseases. Prog Mol Biol Transl Sci. 2009;89:31-95. doi: 10.1016/S1877-1173(09)89003-0. Epub 2009 Oct 7. PMID 20374733
- [Result] Voigt MR, DeLario GT. Perspectives on abdominal organ preservation solutions: a comparative literature review. Prog Transplant. 2013 Dec;23(4):383-91. doi: 10.7182/pit2013100. PMID 24311404
- [Result] Nawrot I, Wozniewicz B, Tolloczko T, Sawicki A, Gorski A, Chudzinski W, Wojtaszek M, Grzesiuk W, Sladowski D, Karwacki J, Zawitkowska T, Szmidt J. Allotransplantation of cultured parathyroid progenitor cells without immunosuppression: clinical results. Transplantation. 2007 Mar 27;83(6):734-40. doi: 10.1097/01.tp.0000258601.17505.9d. PMID 17414706